CLINICAL TRIAL: NCT06878430
Title: Reducing Risk of Stroke and DementIa In patientS With COVert cERebrovascular Disease: a Pilot and Development Study
Brief Title: Reducing Risk of Stroke and DementIa In patientS With COVert cERebrovascular Disease
Acronym: DISCOVER
Status: Not yet recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC25041; HIPS/23/02 (Other Grant/Funding Number: Chief Scientist's Office, Scotland, UK)
Record Dates: First submitted 2025-03-06; First posted 2025-03-17 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Covert Cerebrovascular Disease
Keywords: ccd
MeSH Terms: conditions — Myopathy, Central Core | interventions — Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Functional and Cognitive scores — We will collect information about prior neurological symptoms, including prior symptoms suggestive of TIA or stroke, cognitive or motor symptoms, blood pressure and other known vascular risk factors, medicines, frailty, functional status, education, and employment status We will collect a baseline validated function and cognitive score, and take a sample of speech. Speech will be measured at assessment, in collaboration with the NeuroCARE Clinical and Digital Measures Module (22/SS/0010 IRAS No. 310885).

SUMMARY:
The purpose of the DISCOVER study is to pilot acceptable approaches to people with covert cerebrovascular disease (CCD) and their follow-up. This is the first step in designing efficient randomised trials of treatments to reduce the risk of stroke or dementia in people with CCD.

DETAILED DESCRIPTION:
DISCOVER is a prospective cohort involving individuals with covert cerebrovascular disease (CCD) in NHS Lothian. Participants will be recruited through electronic health records and clinician collaborators. Participants will be monitored at 3 and 6 months and where possible 12 months to assess cognitive, functional, and vascular event outcomes.

ELIGIBILITY:
Inclusion Criteria:

* People who, at the time the letter is prepared or are identified by a clinician

  * Age ≥ 65 years
  * Have no known history of:

    * Stroke or TIA
    * Dementia
    * Parkinson's disease
    * Multiple sclerosis
    * Metastatic cancer (or non-meningioma brain tumour).
  * A CT or MRI scan report ≤5 years before study start date with of one or more of:

    * Cerebral small vessel disease
    * Deep old ischaemic stroke
    * Cortical old ischaemic stroke

Exclusion Criteria:

* Text of brain scan report unreadable
* Do not consent to take part in study procedures
* Unable to consent
* Unable to communicate by email, letter or telephone through language, speech disability or lack of address
* Unlikely to survive one year past enrolment in judgement of the study investigator

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: People aged 65 years or older living in Scotland, UK
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Functional scores | At 3, 6 and 12 months following enrolment
  The investigators will measure day-to-day function with the Bristol Activities of Daily Living Scale, which is a 20-item assessment of daily living abilities for dementia. Each activity has 5 statement options (a - e) which refer to a different level of ability.
Cognitive scores | At 3, 6 and 12 months following enrolment
  The investigators will measure concerns or anxiety about covert cerebrovascular disease using the Montreal Cognitive Assessment. It is a 10-minute test that assesses seven areas of cognition for a total possible score of 30 points. A score of 25 or less is indicative of cognitive impairment.
Speech samples | At 3, 6 and 12 months following enrolment
  Speech will be measured at assessment, in collaboration with the NeuroCARE Clinical and Digital Measures Module (22/SS/0010 IRAS No. 310885).
Vascular events | At 3, 6 and 12 months following enrolment
  At each assessment the investigators will ask about dementia, mild cognitive impairment and stroke symptoms.

IPD SHARING:
Plan to Share IPD: No
Published results will not contain any personal data that could allow identification of individual participants.